CLINICAL TRIAL: NCT06289517
Title: A Study to Evaluate 68Ga-Her2-affibody PET/CT Imaging of Her2 Expression in Tumors
Brief Title: PET Imaging of 68Ga-Her2-affibody in Tumors with High Her2 Expression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Lei YIN, Principal Investigator, Peking University First Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 68Ga-Her2-affibody
Record Dates: First submitted 2024-02-25; First posted 2024-03-04 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Neoplasms
Keywords: 68Ga-Her2-affibody; PET/CT; Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-Her2-affibody (Experimental): Subjects with suspected or confirmed breast cancer will receive an intravenous injection of 68Ga-Her2-affibody followed by PET imaging.
  Interventions: Drug: 68Ga-Her2-affibody

INTERVENTIONS:
Drug: 68Ga-Her2-affibody — 68Ga-Her2-affibody is injected intravenously with a dose of 0.06-0.08 mCi/kg.
  Other Names: Her2 specific PET imaging

SUMMARY:
This project uses HER2 protein as the target group of radiodrugs to explore the diagnostic efficacy, safety and metabolic characteristics of 68Ga-Her2-affibody in the expression status of HER2, aiming to provide a new imaging method for the determination of HER2 status in breast cancer At the same time, it also provides new methods and means for early diagnosis, accurate staging, recurrence judgment, treatment decision-making and prognosis judgment of malignant tumors such as lung cancer, gastrointestinal cancer and bladder cancer, and provides scientific basis for precise treatment of malignant tumors.

DETAILED DESCRIPTION:
This project uses HER2 protein as the target group of radiodrugs to explore the diagnostic efficacy, safety and metabolic characteristics of 68Ga-Her2-affibody in the expression status of HER2 in whole body cancer lesions, aiming to provide a new imaging method for the determination of HER2 status in breast cancer and supplement more overall information that is difficult to obtain by traditional core needle biopsy. At the same time, it also provides new methods and means for early diagnosis, accurate staging, recurrence judgment, treatment decision-making and prognosis judgment of malignant tumors such as lung cancer, gastrointestinal cancer and bladder cancer, and provides scientific basis for precise treatment of malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

- patients with confirmed or suspected cancer; Signed written informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
The diagnostic efficacy of 68Ga-Her2-affibody PET/CT in the evaluation of breast cancer | 1 year
  the standardized Uptake Value (SUV) of lesions on 68Ga-Her2-affibody PET/CT

SECONDARY OUTCOMES:
The dosimetry of 68Ga-Her2-affibody | 1 year
  Research on the dose distribution of 68Ga-Her2-affibody in cancer patients by 1-hour dynamic PET/CT acquisition and analyze by the dosimetry software
Quantitative evaluation of 68Ga-Her2-affibody | 1 year
  Analyze Her2 expression at the imaging level in combination with Her2 expression
Correlation with pathological expression | 1 year
  Analyze Her2 expression at the imaging level in combination with Her2 expression in pathological specimens

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao Y, Yin L, Duan X, Fu Z, Liu Q, Chen J, Xin L, Zhu X, Xiang H, Xu L, Ye J, Liu M. HER2-targeted PET/CT imaging provides potential biomarkers for differentiating HER2-zero, -low, and -positive breast cancer. Eur J Nucl Med Mol Imaging. 2025 Oct;52(12):4525-4538. doi: 10.1007/s00259-025-07220-3. Epub 2025 May 8. PMID 40338302